CLINICAL TRIAL: NCT02875561
Title: A Randomized Controlled Trial of Ultrasonic Aspiration Versus CO2 Laser Ablation for the Treatment of Vulvar Intraepithelial Neoplasia
Brief Title: Ultrasonic Aspiration Versus CO2 Laser Ablation for the Treatment of Vulvar Intraepithelial Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Stryker Instruments (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0701.cc
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Vulvar Intraepithelial Neoplasia (VIN)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sonopet Ultrasonic Aspirator (Active Comparator): Treatment of VIN dysplasia with sonopet ultrasonic aspirator: to evaluate the incident of recurrence of VIN dysplasia events in women treated for VIN with the sonopet ultrasonic aspirator compared to CO2 Laser Ablation
  Interventions: Device: Sonopet Ultrasonic Aspirator
- CO2 Laser Ablation (Experimental): Treatment of VIN dysplasia with CO2 Laser Ablation: to evaluate the incident of recurrence of VIN dysplasia events in women treated for VIN with the sonopet ultrasonic aspirator compared to CO2 Laser Ablation
  Interventions: Device: CO2 Laser Ablation

INTERVENTIONS:
Device: Sonopet Ultrasonic Aspirator — To evaluate the incident of recurrence of VIN dysplasia events in women treated for VIN with the sonopet ultrasonic aspirator compared to CO2 Laser Ablation
  Arms: Sonopet Ultrasonic Aspirator
Device: CO2 Laser Ablation — To evaluate the incident of recurrence of VIN dysplasia events in women treated for VIN with the sonopet ultrasonic aspirator compared to CO2 Laser Ablation
  Arms: CO2 Laser Ablation

SUMMARY:
The primary objective of this study is to evaluate the incidence of vulva dysplasia recurrence within 12 months of treatment with Carbon Dioxide (CO2) laser ablation or ultrasonic aspiration.

DETAILED DESCRIPTION:
Incidence of Vulvar Intraepithelial Neoplasia (VIN) is increasing among women and there still lacks a standard of care for optimal treatment. Current treatment options aim to treat the symptoms associated with VIN and result in a high recurrence rate. Due to the high reoccurrence rate and the nature of the current treatments, a more effective treatment option is warranted. An effective treatment that targets only the diseased areas could potentially decrease recurrence rates. Additionally, a more conservative treatment modality could contribute to reduced risks of scarring, discomfort, and psychosocial and sexual distraught. The researchers hypothesize that treatment for VIN with ultrasonic aspiration will have a 60% reduction in recurrence rates over 12 months as compared to CO2 laser aspiration.

This study will employ a randomized controlled trial (RCT) design. This is a phase III study to determine the effectiveness of a more targeted treatment therapy for VIN (comparing ultrasonic aspiration versus CO2 laser ablation). Potential participants will be identified through the gynecological clinical practices following diagnosis of high grade VIN and will be randomized (1:1) to one of the treatment therapies. Randomization will be stratified for multi-focal disease and Human Papillomavirus (HPV) status. Both the Sonopet Ultrasonic Aspirator and the CO2 laser ablation devices are FDA approved devices for the treatment of vulvar dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-89 years old
* Women diagnosed with high-grade VIN (diagnosed by pathology)
* Women referred for vulva sparing treatment for dysplasia
* Women available for follow-up of treatment for 12 months

Exclusion Criteria:

* Women who are pregnant
* Women with low-grade VIN dysplasia (diagnosed by pathology)
* Women with vaginal intraepithelial neoplasia(VAIN)
* Women requiring vulvectomy for treatment
* Women unable to provide informed consent

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-03-26 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saketh Guntupalli, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - University of Oklahoma, Norman, Oklahoma

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sonopet Ultrasonic Aspirator | CO2 Laser Ablation
Started | 19 | 28
Completed | 19 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sonopet Ultrasonic Aspirator | CO2 Laser Ablation | Total
Number analyzed (Participants) | 19 | 28 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 34
  >=65 years | 3 | 10 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 28 | 47
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 27 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 28 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence of Dysplasia
Description: Number of participants with recurrence of dysplasia time point 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sonopet Ultrasonic Aspirator | CO2 Laser Ablation
Number analyzed (Participants) | 19 | 28
Participants | 5 | 8

2. Secondary Outcome: Number of Participants With Scarring
Description: Physical evaluation for scarring
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sonopet Ultrasonic Aspirator | CO2 Laser Ablation
Number analyzed (Participants) | 19 | 28
Participants | 6 | 12

3. Secondary Outcome: Changes in Sexual Function
Description: Evaluated by Female Sexual Function Index Scale Title: Female Sexual Function Index (FSFI) Minimum value: 2.0 Maximum value: 36.0 a score of 0 in any domain correlates to no sexual activity. a score of 0 in any domain correlates to no sexual activity in that domain alone, and is not indicative of the total score. Lower scores indicate worse sexual function.
Time Frame: Baseline (enrollment), 12 months
Population: all surveys at all timepoints were optional. Some participants completed all surveys, some completed only baseline surveys and some only completed end of study surveys. This is why the population varies between timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sonopet Ultrasonic Aspirator | CO2 Laser Ablation
Number analyzed (Participants) | 15 | 24
score on a scale
  Baseline | 14.9 (12.3) | 10.9 (9.5)
  End of Study: number analyzed (Participants) | 8 | 11
  End of Study | 10.3 (11.3) | 19.8 (10.1)

4. Secondary Outcome: Changes in Mental and Physical Wellness
Description: Evaluated by Functional Assessment of Cancer Therapy - Vulva (FACT-V) health survey for vulva disease Scale Title: Functional Assessment of Cancer Therapy - Vulva (FACT-V) High score correlates to better quality of life. This survey uses a 5-point Likert type scale. Minimum score: 0 Maximum score: 184
Time Frame: Baseline (enrollment), End of Study (12 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sonopet Ultrasonic Aspirator | CO2 Laser Ablation
Number analyzed (Participants) | 16 | 25
score on a scale
  Baseline | 155.6 (29.8) | 145 (29.1)
  End of Study: number analyzed (Participants) | 9 | 11
  End of Study | 147 (26.4) | 156.5 (20.9)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Sonopet Ultrasonic Aspirator | CO2 Laser Ablation
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/28
Other Adverse Events (participants affected / at risk) | 12/19 | 18/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sonopet Ultrasonic Aspirator (N=19) | CO2 Laser Ablation (N=28)
discomfort (General disorders) | 1 (1) | 2 (2)
pain (General disorders) | 4 (4) | 4 (4)
vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 3 (3)
discharge (Reproductive system and breast disorders) | 3 (3) | 1 (1)
anal pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
tenderness (General disorders) | 1 (1) | 2 (2)
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
infection (Infections and infestations) | 0 (0) | 1 (1)
irritation (General disorders) | 1 (1) | 1 (1)
yeast infection (Infections and infestations) | 0 (0) | 1 (1)
itching (General disorders) | 1 (1) | 1 (1)
soreness at site (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT02875561/Prot_SAP_000.pdf